CLINICAL TRIAL: NCT07275632
Title: A Multicenter, Single-Arm, Exploratory Study Evaluating the Effect of Perioperative Oral Vonoprazan Fumarate on the Incidence of Delayed Graft Function in Deceased Donor Kidney Transplant Recipients
Brief Title: The Effects of Vonoprazan Fumarate on DGF Incidence in DD Kidney Transplant Recipients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Weiyang He, Professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZZ2025-945-01
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Delayed Graft Function; Kidney Transplantation
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vonoprazan Fumarate (Experimental)
  Interventions: Drug: Vonoprazan fumarate

INTERVENTIONS:
Drug: Vonoprazan fumarate — Phase Ib:
  A dose escalation study will be initiated with vonoprazan fumarate 20 mg once daily (qd). Two dose groups are planned: 20 mg qd and 20 mg twice daily (bid). According to a "3+3" dose escalation scheme, the first three subjects will receive vonoprazan fumarate 20 mg qd orally, starting on the day of kidney transplantation and continuing until postoperative day 7. Safety and tolerability will be assessed from the day of transplantation through postoperative days 7 and 28.
  Phase II:
  An expansion study will be conducted at the recommended Phase II dose of vonoprazan fumarate to evaluate the efficacy, safety, and tolerability of the regimen. Vonoprazan fumarate will be administered orally, starting on the day of kidney transplantation and continuing daily until postoperative day 7.
  Throughout both the Phase Ib and Phase II stages, all recipients will receive the center's standard immunosuppressive regimen.

SUMMARY:
This is an exploratory, multicenter, single-arm study designed to evaluate the efficacy of perioperative Vonoprazan Fumarate in reducing the incidence of Delayed Graft Function (DGF) in deceased-donor kidney transplant recipients. DGF is a common early complication that significantly impacts graft function and long-term transplant survival. This study aims to explore how Vonoprazan Fumarate, a potassium-competitive acid blocker (P-CAB), can potentially improve macrophage phagocytic function, reduce kidney inflammation, and enhance early kidney function recovery.

Patients aged 18 years and older who are undergoing first-time deceased-donor kidney transplantation will be enrolled. Vonoprazan Fumarate will be administered daily starting on the day of transplantation and continuing for seven days post-surgery. The primary endpoint is DGF incidence, while secondary endpoints include kidney function recovery, serum creatinine reduction, estimated glomerular filtration rate, and safety assessments. Adverse events will be monitored, and the study will also explore potential biomarkers for inflammation and graft function.

The study is expected to provide insights into a potential new therapeutic strategy to reduce DGF and improve early kidney transplant outcomes, potentially benefiting future kidney transplant patients by offering a safer and more effective perioperative treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of transplantation.
* Undergoing first-time deceased-donor kidney transplantation.
* No administration of proton-competitive acid blockers (P-CABs) in the 1 month prior to transplantation.
* Consent to receive the standard immunosuppressive therapy post-transplantation.
* Ability and willingness to provide informed consent and comply with study procedures and follow-up.
* Complete baseline clinical data available.

Exclusion Criteria:

* Receiving a living-donor kidney transplant or multi-organ transplantation.
* Previous history of any solid organ or cellular transplantation (with the exception of corneal transplants).
* Intraoperative occurrence of hyperacute rejection or confirmed graft non-function (e.g., renal artery thrombosis).
* Presence of high risk for primary graft non-function (e.g., severe injury to the transplant renal artery).
* Severe postoperative intestinal obstruction requiring prolonged fasting or inability to take oral medication in perioperative period.
* Known history of hypersensitivity to vonoprazan fumarate or any of its excipients.
* Subjects with severe hepatic impairment (Child-Pugh Class C).
* Concomitant use of strong CYP3A4 inhibitors (e.g., ritonavir, clarithromycin).
* Current therapy with atazanavir or rilpivirine.
* Any other condition deemed by the investigator to be inappropriate for study participation (e.g., uncontrolled active infection, severe peptic ulcer, pregnancy or lactation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Delayed Graft Function (DGF) | Within the first 7 days post-transplant
  Delayed Graft Function (DGF) is defined as the requirement for any form of dialysis (hemodialysis or peritoneal dialysis) due to renal insufficiency within the first week after kidney transplantation.

SECONDARY OUTCOMES:
The rate of serum creatinine decline | Postoperative days 1 to 7
  The rate of serum creatinine decline will be calculated on a daily basis from postoperative day 1 to day 7.
Estimated Glomerular Filtration Rate (eGFR) | Postoperative days 1 to 7
  eGFR will be measured daily from postoperative day 1 through day 7.
Daily urinary output | Postoperative days 1 to 7
  Daily urinary output will be recorded from postoperative day 1 through day 7.
Incidence of Adverse Events | Fecal routine tests will be performed on postoperative days 3 and 7. All other AEs will be monitored daily during the first 7 postoperative days.
  Adverse events-specifically renal (e.g., acute rejection), gastrointestinal (e.g., bloody stools, acid reflux), and electrolyte imbalance (e.g., hypomagnesemia, hyperkalemia)-will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou

IPD SHARING:
Plan to Share IPD: No